CLINICAL TRIAL: NCT01030198
Title: Post-Market, Two-Arm, Single Blind, Controlled Study of the RevLite Electro-optic Q-Switched Neodymium-doped Yttrium Aluminum Garnet (EO QS Nd:YAG) Laser System for the Treatment of Scars
Brief Title: Laser Treatment for Fresh Surgical Scars and Mature Scars
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C68-08-S
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: New Surgical Scars; Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fresh surgical scars (Experimental): Treatment of scars
  Interventions: Device: RevLite (Laser Treatment)
- Mature scars (Experimental): Treatment of scars
  Interventions: Device: RevLite (Laser Treatment)

INTERVENTIONS:
Device: RevLite (Laser Treatment)

SUMMARY:
The purpose of this study is to measure the effectiveness of the RevLite Laser in the treatment of both fresh surgical scars and mature/older scars.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I-VI and either a fresh surgical scar (with sutures still present [or dissolving sutures within 7 days of surgery for facial scars or within 14 days of surgery for scars on the trunk or extremities) of at least 2cm in length or an erythematous and/or hypertrophic scar of at least 2cm in length and of greater than or equal to 18 months in duration
* Scar is easily divisible into two equal segments for the purpose of the study, or is bilateral in nature (e.g., inframammary)

Exclusion Criteria:

* Pregnant, lactating, or is planning to become pregnant
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* any skin pathology/condition that could interfere with evaluation or requires the use of interfering topical systemic therapy
* coagulation disorder or currently using anti-coagulation medication (including but not limited to heavy aspirin therapy)
* any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in the study
* currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 30 days
* unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function
* unreliable for the study, including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits
* Isotretinoin therapy within 6 months
* need to be exposed to artificial tanning devices or excessive sunlight during the trial
* prior treatment with parenteral gold therapy
* does not agree to refrain from other laser treatment, (micro)dermabrasion or topical scar treatment creams for the duration of the study
* Diabetes Type 1 or 2
* Lupus, scleroderma or similar immune system disorder
* underlying silicone or other non-absorbable filler in the area of the scar
* phenol chemical peel or dermabrasion to the area of the scar within 3 months
* Fitzpatrick Skin Type IV, V or VI with a known sensitivity to hydroquinone or is unwilling or unable to comply with physician/manufacturer instructions for the use of this ingredient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sanctuary Medical Aesthetic Center, Boca Raton, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fresh Surgical Scars; Mature Scars: Device: RevLite (Laser Treatment)
Period: Overall Study
Arm/Group | Fresh Surgical Scars | Mature Scars
Started | 0 (None recruited) | 7
Completed | 0 (None recruited) | 0 (Study terminated due to poor results and lack of enrollment)
Not Completed | 0 | 7
Not completed — Could not measure efficacy accurately | 0 | 7

BASELINE CHARACTERISTICS:
Population: There were no baseline participants who were analyzed that had fresh surgical scars. This study was not completed due to the lack of enrollment.
Groups:
- Fresh Surgical Scars; Mature Scars: Treatment of scars
  Device: Revlite
- Total: Total of all reporting groups
Arm/Group | Fresh Surgical Scars | Mature Scars | Total
Number analyzed (Participants) | 0 | 7 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 7 | 7
  >=65 years |  | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 48.4 (10.2) | 48.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 7 | 7
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Improvement in Scar Appearance, Vascularity, Height, Pliability, Pigmentation and Any Pre-existing Pruritis
Description: The number of participants who experienced improvements in scar appearance, vascularity, height, pliability, pigmentation and any pre-existing pruritis will be counted.
Time Frame: 1 month post final treatment (fresh scars) or 3 and 6 months post final treatment (mature scars)
Population: Could not measure accurately with measurement tools.
Groups:
- Fresh Surgical Scars; Mature Scars: Treatment of scars
  RevLite (Laser Treatment)
Arm/Group | Fresh Surgical Scars | Mature Scars
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events occurring were captured and followed until the study was terminated, approximately 11 months.
Description: The number of patients at risk is zero because no patients were enrolled in the fresh surgical study arm.
Arm/Group | Fresh Surgical Scars | Mature Scars
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/7
Other Adverse Events (participants affected / at risk) | 0/0 | 0/7

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.